CLINICAL TRIAL: NCT00690105
Title: Comparative, Multicentre, Randomized, Double-blind Study to Assess the Efficacy of Tacrolimus 0.1% Ointment Versus Fluticasone 0.005% Ointment in Adult Patients Suffering From Moderate to Severe Atopic Dermatitis and Presenting With So-called 'Red Face' Lesions of the Head and Neck.
Brief Title: Protopic Ointment in Adult Atopic Eczema of the Face
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FG-506-06-FR-04; EUDRACT #: 2004-002477-23
Record Dates: First submitted 2008-06-02; First posted 2008-06-04 (Estimated); Last update posted 2014-09-01 (Estimated); Status verified 2014-08

CONDITIONS: Dermatitis, Atopic
Keywords: Dermatitis, Atopic; Dermatologic Agents; Topical Drug Administration; Tacrolimus; Calcineurin; Corticosteroid; Fluticasone propionate; Face
MeSH Terms: conditions — Dermatitis, Atopic; Facies

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental)
  Interventions: Drug: tacrolimus 0.1%
- B (Active Comparator)
  Interventions: Drug: fluticasone 0.005 %

INTERVENTIONS:
Drug: tacrolimus 0.1% — ointment
  Other Names: Protopic® 0.1%
  Arms: A
Drug: fluticasone 0.005 % — ointment
  Other Names: Flixovate® 0.005%
  Arms: B

SUMMARY:
Patients with facial atopic eczema and a poor response to topical corticosteroid applied either Protopic or Fluticasone ointment twice a day for 3 weeks. They could continue during 3 more weeks once a day if needed or change for the other ointment.

DETAILED DESCRIPTION:
Treatments were to be applied twice daily over all lesions on the face (except for the eyelids) until clearance, for a maximum of 3 weeks and then, in case of uncleared residual lesions, once daily for up to 3 further weeks. In the event of a flare-up the treatment was to be resumed twice a day until the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe AD (Rajka & Langeland score) with lesions to the head and neck defined as 'red face' or 'facial eczema': erythema affecting at least 10% of the surface of the 'face' (head, neck, chest, nape of neck), due to long-term AD
* At least two flare-ups of 'facial' eczema during the 12 months prior to inclusion and, in the investigator's opinion, conventional treatment had proved ineffective or poorly tolerated
* Female patients of childbearing age: effective means of contraception throughout the period of the study and for four weeks following the end of the study
* Informed consent
* Therapeutic washout for atopic dermatitis treatments

Exclusion Criteria:

* Genetic epidermal barrier defect, such as Netherton's syndrome, or suffering from erythroderma
* Seborrheic dermatitis or contact dermatitis affecting the 'face', or any other facial erythema of non-atopic origin
* Clinical infection due to the VZV virus (varicella, zona), HSV1-2 viruses (herpes), verruca vulgaris or molluscum contagiosum
* Superinfected eczema
* Known hypersensitivity to macrolides or to any other excipient in tacrolimus 0.1% ointment
* Known hypersensitivity to one of the agents contained in the fluticasone 0.005% ointment preparation
* Ulcerated lesions, of whatever type
* Moderate to severe acne or rosacea
* Patients who participated at the same time in another clinical study or who had participated in another clinical study within 28 days prior to inclusion in the study
* Any type of substance abuse (including that of drugs and alcohol) or any mental disorder/psychological state which, in the investigator's opinion, might interfere with the patient's follow-up
* Serologically-proven HIV positivity

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 577 (Actual)
Dates: Start 2004-02; Primary Completion 2005-07 (Actual); Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
Percentage of patients presenting at the week 3 visit (day 21) with an improvement of at least 60% in their local mEASI score (mLEASI) compared to Baseline (day 1). | 3 weeks

SECONDARY OUTCOMES:
Percentage of patients no longer presenting with 'facial' erythema at day 7 and day 21 | 1 week and 3 weeks
Assessment of facial pruritus at day 1, day 7 and day 21 | 1 week and 3 weeks
Global assessment of clinical response on the 'face' by the physician at day 7 and day 21 | 1 week and 3 weeks
Global assessment of clinical response on the 'face' by the patient at day 7 and day 21 | 1 week and 3 weeks
Patient's quality of life at day 1 and day 21 | 1 week and 3 weeks
mLEASI score values at day 7 and day 21 | 1 week and 3 weeks
Physician's assessment of individual signs | 1 week and 3 weeks
Quality of sleep at day 1, day 7 and day 21 | 1 week and 3 weeks
Affected surface area assessment at day 1, day 7 and day 21 | 1 week and 3 weeks
Number of patients using the ointment from the other group to treat facial lesions after day 21 | 3 weeks
Incidences of adverse events during the study period | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Central Contact, Study Director — Astellas Pharma Europe B.V.
Locations (1):
- Nice, France